CLINICAL TRIAL: NCT06944002
Title: The Effect of Milk Consumption on the Blood Microbiome in Healthy Volunteers
Brief Title: Milk Consumption and Blood Microbiome in Healthy Volunteers
Acronym: MAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: NWO (Dutch Organisation for Scientific Research) (Unknown)
Responsible Party: Principal Investigator, Maikel Petrus Peppelenbosch, prof. dr, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL88008.078.24; KICH2.V4P.22.015 (Other: NWO (Dutch organisation for scientific research))
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: The blood microbiome; The gut microbiome; Milk consumption; Healthy volunteers
MeSH Terms: interventions — Cultured Milk Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Milk consumption (Experimental): Milk consumption for 7 days
  Interventions: Dietary Supplement: Milk product

INTERVENTIONS:
Dietary Supplement: Milk product — The participants will abstain from consumption of any dairy product for ten days and subsequently drink milk for seven consecutive days (700 ml per day), while concomitant consumption of other dairy products is also allowed.

SUMMARY:
The goal of this study is to learn if cfDNA of milk-associated intestinal bacteria (MAIB) is detectable in the bloodstream. The primary question it aims to answer is:

- Does milk consumption simultaneously increase the number of MAIB cfDNA counts in blood samples, as it does in fecal samples?

Researchers will compare cfDNA counts of MAIB to those of fecal samples to assess whether the blood microbiome is a valid measure of the gut microbiome, utilizing a self-developed bioinformatics pipeline.

Participants will:

* Abstain from consuming any dairy products for ten days, followed by drinking milk for 7 consecutive days.
* Provide blood and fecal samples before dairy abstinence, as well as at 0, 24, and 48 hours, and one week after the reintroduction of milk.

DETAILED DESCRIPTION:
eDNA (ecological DNA) is a concept that is gaining popularity for making comprehensive descriptions of all organisms present in an ecosystem. Gut microbiomes can be considered a specific variant of eDNA. In theory, a description of the gut microbiome should contain all different kinds of microorganisms in our gastrointestinal tract, including bacteria, viruses, archaea, fungi and other organisms (e.g. worms and phages). In practice, making such descriptions is challenging because of spurious temporal changes and technical challenges (e.g. the commonly used 16S rRNA approach ignores many organisms). Nevertheless, making accurate descriptions is essential as it is generally accepted that the gut microbiome plays critical roles in maintaining host homeostasis and health.

To overcome the challenges in sampling the intestinal microbiome, most investigators currently rely on probing faeces. We have pioneered the field in developing improved technical approaches; for example, we previously performed a double-balloon endoscopic study in healthy volunteers to characterize this microbiome in its entirety. Problems with the faecal microbiome include its poor capture of the adherent flora (which seems the most relevant concerning human physiology), it is highly heterogeneous and can cause results to differ depending on which part of faecal samples was taken, and technological challenges, as many eukaryotes are quite resistant to DNA isolation protocols. Additionally, the faecal microbiome is dominated by diet, which can vary substantially from day to day in humans. For example, faecal material deriving from breakfast can have a significantly different microbiological composition compared to that derived from dinner. Hence, there is a call for alternatives.

The blood microbiome is a newly discovered way of probing the microbiome, integrating the colonization of all kinds of body sites, particularly the intestinal tract. It is speculated that the DNA fragments of various microorganisms enter the circulation through mechanisms that are yet fully understood. The gastrointestinal microbiome is considered a major source of blood microbiome, especially in the case of an impaired gut barrier, which can occur in various chronic diseases.

The description of the entire body of cell-free DNA fragments that derive from non-human origin is called the blood microbiome, even though it does not constitute living organisms, but rather their remnants. The blood microbiome signature has been reported as a predictable biomarker in differentiating patients with cancer from healthy individuals and even for distinguishing between different cancer types. However, the approach remains very controversial due to bioinformatical pitfalls. While we have invested substantial energy in resolving the issues involved, the field requires a formal proof-of-concept to progress. The current study is meant to provide this.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* 18.5 =< BMI < 25 kg/m2
* All genders included
* Not be lactose intolerant
* Willing to consume milk

Exclusion Criteria:

* Regularly used medications such as antibiotics, steroids, beta blockers, and adrenergic- stimulating agents (self-report)
* Regular use of prebiotic and/or probiotics apart from yogurt and young soft cheese (self-report)
* Antibiotic intake in the previous months (self-report)
* Daily consumption of more than 10 cigarettes (self-report)
* Chronic diseases including type 2 diabetes, hypertension, fatty liver disease, cancer, or autoimmune disease (self-report)
* Internal diseases, including those of the gastrointestinal tract, lung, heart, vasculature, liver, and kidney (self-report)
* Eating disorder or unconventional eating habits (self-report)
* Participation in another study (self-report)
* Women: pregnancy and breastfeeding (self-report)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Lactococcus DNA counts | 10 days before milk consmuption (baseline), 0, 1, 2 and 7 days during milk consumption
  Changes in blood and fecal Lactococcus DNA during milk consumption will be measured with shotgun sequencing technology.

SECONDARY OUTCOMES:
Changes in other microbial DNA counts | 10 days before milk consmuption, 0, 1, 2 and 7 days during milk consumption
  Changes in other blood and fecal microbial DNA counts during milk consumption will be measured with shotgun sequencing technology.

OTHER OUTCOMES:
Change in BMI | 10 days before milk consmuption, 0, 1, 2 and 7 days during milk consumption
  Weight in kilograms and height in meters will be combined to report BMI in kg/m^2.
Change in systolic and diastolic blood pressure | 10 days before milk consmuption, 0, 1, 2 and 7 days during milk consumption
  Changes in both systolic and diastolic blood pressure during milk consumption will be assessed with a blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Maikel P Peppelenbosch, MD, PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus MC - Department of Gastroenterology and Hepatology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anomised IPD used in the results of the publication will be shared in full
Supporting Information: Study Protocol
Time Frame: from appearance of the study on the preprint server to at least January 20, 2035
Access Criteria: the anomised data will be available to everyone
URL: https://www.eur.nl/en/library/research-support/eur-data-repository

REFERENCES:
- [Derived] Su J, Hansen BE, Wang Z, Sharmenov A, Xia X, Broekhuizen M, Ma Z, Peppelenbosch MP. Yogurt reintroduction and the circulating microbiome in healthy volunteers: protocol for a prospective, longitudinal, species-controlled crossover clinical trial (MAMI). Contemp Clin Trials Commun. 2025 Nov 24;48:101579. doi: 10.1016/j.conctc.2025.101579. eCollection 2025 Dec. PMID 41399631